CLINICAL TRIAL: NCT07359963
Title: An Exploratory Clinical Study on the Intravenous Infusion of REGEND007 (Generic Airway Basal Layer Stem Cell Preparation) for the Treatment of Idiopathic Pulmonary Fibrosis (IPF).
Brief Title: Treatment of Idiopathic Pulmonary Fibrosis (IPF) by REGEND007 Cell Therapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REGEND007-IPF-251
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGEND007 Cell Therapy (Experimental)
  Interventions: Biological: REGEND007 Cell Therapy

INTERVENTIONS:
Biological: REGEND007 Cell Therapy — This study's intravenous infusion dose escalation protocol is based on a 3+3 dose escalation design, with a total of 4 dose groups. Each group included 3 subjects, and the dose is gradually increased until the maximum tolerated dose(MTD) or the maximum administered dose (MAD) is reached.

SUMMARY:
This study is a prospective, single-arm, dose-escalation exploratory clinical trial to investigate the safety, tolerability and preliminary efficacy of REGEND007 stem cell preparation administered by intravenous infusion in the treatment of idiopathic pulmonary fibrosis (IPF), with a follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Gender is not restricted. When signing the informed consent form, the age should be between 40 and 80 years old (inclusive of the boundary value).
* Diagnosed with idiopathic pulmonary fibrosis (IPF).
* During the screening process, the six-minute walk test should be ≥ 150 meters and < 600 meters; or the lung function FVC should be > 30% of the predicted value.
* Voluntarily sign the informed consent form, be able to cooperate with the completion of research-related procedures and examinations, and be able to comprehensively describe or record the changes in the condition.

Exclusion Criteria:

* Female subjects who are pregnant, breastfeeding, or planning to become pregnant within one year after using this product; or male subjects whose partner is planning to become pregnant.
* Subjects selected during the screening whose estimated survival period is less than one year.
* Subjects selected during the screening who have a current or past history of malignant tumors (excluding malignant tumors with a disease-free survival of more than five years and judged by the researcher to have a relatively mild invasiveness, such as non-melanoma skin cancer, invasive cervical cancer, bladder cancer, thyroid cancer, and breast cancer, etc.).
* Subjects selected within 4 weeks before diagnosis of pneumonia (including bacterial, fungal or viral pneumonia).
* Subjects selected within 4 weeks before an acute exacerbation of IPF.
* Subjects selected within 4 weeks before having one or more results reported by pathogenological or serological tests (nucleic acid, antigen, virus culture, specific IgG antibody levels) indicating novel coronavirus infection, or suspected novel coronavirus infection (manifesting symptoms such as fever, headache, fatigue, joint pain, runny nose, sore throat, and persistent cough, and the disease course is consistent with the prevalent strain).
* Subjects selected within 4 weeks before having a history of invasive or non-invasive mechanical ventilation.
* Subjects selected during the screening who have active pulmonary tuberculosis, poorly controlled bronchial asthma, acute pulmonary embolism, severe pulmonary hypertension [cardiac ultrasound examination > 70 mmHg], etc.
* Subjects selected within 6 months before having a serious non-pulmonary systemic disease and judged by the researcher as not suitable to participate in this study, such as diabetes with ketoacidosis or hyperosmolar coma, acute myocardial infarction, unstable angina pectoris, NYHA heart failure grade III/IV, stroke, liver cirrhosis with severe liver dysfunction, severe renal insufficiency, etc.
* Subjects selected during the screening who have severe anemia, or controlled poorly granulocytopenia or thrombocytopenia.
* Subjects selected during the screening who have a history of suicide risk, psychiatric history or epilepsy history.
* Subjects selected during the screening who have severe malnutrition.
* Subjects selected during the screening whose 12-lead electrocardiogram shows severe arrhythmias (such as ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or second-degree and above conduction abnormalities of the heart.
* Subjects selected within 4 weeks before participating in other clinical trials with intervention measures or using other biological agents for treatment.
* Researchers, collaborating researchers, research coordinators, researchers participating in the study or employees of the research center or their family members.
* Subjects selected during the screening who the researcher considers unsuitable to participate in the trial (increasing the risk for the subjects or interfering with the clinical trial).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of drug-related adverse events (AEs) | 12 weeks after the administration
  All adverse medical events that occur from the time the subject signs the informed consent form. These can manifest as symptoms, signs, diseases, or abnormal laboratory test results, but they do not necessarily have a causal relationship with the investigational drug.

SECONDARY OUTCOMES:
The change in the actual forced vital capacity (FVC) compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration
  FVC is the full amount of air that can be-exhaled with effort in a complete breath
The change in forced vital capacity (FVC) actual-to-predicted ratio compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  The FVC actual-to-predicted ratio is a crucial indicator in pulmonary function tests, and it is mainly used to determine whether there is restrictive ventilation dysfunction.
The change in the actual forced expiratory volume in one second (FEV1) compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration
  FEV1 is the volume of breath exhaled with effort in one second.
The change in the forced expiratory volume in one second (FEV1) actual-to-predicted ratio compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration
  The FEV1 actual-to-predicted ratio is a crucial indicator in pulmonary function tests, representing the percentage relationship between the actual measured value of the first-second forced expiratory volume (FEV1) and the predicted value calculated based on individual characteristics. Under normal circumstances, the actual measured value of FEV1 should reach more than 80% of the predicted value.
The change in the carbon monoxide diffusion capacity (DLCO) compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration
  DLCO is a measure of the conductance of CO across the alveolar-capillary membrane and its binding with hemoglobin.
The change in carbon monoxide diffusion capacity (DLCO) actual-to-predicted ratio compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  DLCO actual-to-predicted ratio is a crucial indicator in pulmonary function testing, used to assess the oxygen exchange capacity and efficiency of the alveoli.
The change in the ratio of carbon monoxide diffusion capacity to lung alveolar volume (DLCO/VA) compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  DLCO/VA is also known as the diffusion constant, since the diffusion amount is affected by the alveolar ventilation volume, a decrease in alveolar ventilation volume can lead to a reduction in DLCO. Therefore, this value is often used for correction to eliminate the influence of lung volume on the diffusion amount.
The change in the six-minute walk test (6MWT) compared to the baseline | 24 hours after administration, 4 and 12 weeks after the last administration.
  6MWT is one of the commonly used methods in clinical practice for assessing a patient's cardiac and pulmonary functions, which involves measuring the distance that a patient can walk quickly on a flat and hard surface within 6 minutes.
The time when the first acute exacerbation of IPF occurred after administration | Within 12 weeks after administration
  The time when the first acute exacerbation of IPF occurred after administration is helpful for assessing disease progression and prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No